CLINICAL TRIAL: NCT07060222
Title: Intestinal Preparation in Colonoscopy: Lactulose vs Sodium Phosphate, a Multicenter, Randomized, Double-Blind Comparative Clinical Trial.
Brief Title: Intestinal Preparation in Colonoscopy: Lactulose vs Sodium Phosphate.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Roberto Ulises Cruz Neri, Coloproctologist, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 131/25
Record Dates: First submitted 2025-06-11; First posted 2025-07-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Bowel Preparation for Colonoscopy
Keywords: lactulose; Colonoscopy; sodium phosphate; bowel preparation

STUDY DESIGN:
Intervention Model Description: Multicenter single-blind randomized clinical trial study.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intestinal preparation using sodium phosphate (Active Comparator): Patients will be randomized and assigned a bowel preparation on the day they are given their colonoscopy appointment date.
  Interventions: Combination Product: Bowel preparation before colonoscopy: Sodium phosphate.
- Bowel preparation with lactulose (Active Comparator): Patients will be randomized and assigned a bowel preparation on the day they are given their colonoscopy appointment date.
  Interventions: Combination Product: Bowel preparation before colonoscopy: Lactulose.

INTERVENTIONS:
Combination Product: Bowel preparation before colonoscopy: Lactulose. — In this randomized, multicenter, single-blind clinical trial, each patient who meets our inclusion criteria will be assigned a randomized code to be included in one of the two study arms, that is, one of the groups and the assigned bowel preparation for the colonoscopy. The benefits and minimal risks of participation will be explained to them, and they will also be asked to sign an informed consent form so that we can proceed with the colonoscopy and collect all the necessary data for our protocol and variable analysis.
  Arms: Bowel preparation with lactulose
Combination Product: Bowel preparation before colonoscopy: Sodium phosphate. — In this randomized, multicenter, single-blind clinical trial, each patient who meets our inclusion criteria will be assigned a randomized code to be included in one of the two study arms, that is, one of the groups and the assigned bowel preparation for the colonoscopy. The benefits and minimal risks of participation will be explained to them, and they will also be asked to sign an informed consent form so that we can proceed with the colonoscopy and collect all the necessary data for our protocol and variable analysis.
  Arms: Intestinal preparation using sodium phosphate

SUMMARY:
To compare intestinal preparation with Lactulose vs. Sodium Phosphate as the better agent for performing high-quality colonoscopies at the Civil Hospital Fray Antonio Alcalde and the Civil Hospital Juan I. Menchaca, both in Guadalajara, Mexico; as well as Hospital Santo Tomás in Panama City, Panama; and Hospital Gustavo Nelson Collado Ríos in Chitré, Panama; during the period from April 1, 2025, to November 30, 2025. The comparison will focus on colonoscopy quality, patient tolerance, satisfaction, and electrolyte changes, using the agents orally as part of the bowel preparation prior to the colonoscopy procedure.

DETAILED DESCRIPTION:
Randomized Double-Blind Clinical Trial conducted from April 1, 2025, to November 30, 2025, involving patients scheduled for outpatient colonoscopy at the Coloproctology Departments of the Civil Hospital Fray Antonio Alcalde, Civil Hospital Juan I. Menchaca (both in Guadalajara, Mexico), Hospital Santo Tomás in Panama City, Panama, and Hospital Gustavo Nelson Collado Ríos in Chitré, Panama.

Patients undergoing elective or emergency therapeutic colonoscopies, as well as those with certain medical conditions or pregnancy, were excluded from the study. Factors related to bowel preparation were considered, with particular emphasis on the characteristics of the chosen preparation agent, its effects, and findings observed during each patient's colonoscopy. All data were collected in a database, which will be shared via a digital platform using the SPSS statistical package for data analysis, followed by the development of conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Indication for Scheduled Colonoscopy: Participants must have a valid clinical indication for undergoing a scheduled colonoscopy, such as part of a colorectal cancer screening program, evaluation of gastrointestinal symptoms, or follow-up of previously diagnosed colorectal conditions.
* Ability to Provide Informed Consent: Participants must have the physical and mental capacity to understand the nature of the study and voluntarily provide informed consent to participate.

Exclusion Criteria:

* History of Intestinal Obstruction: Participants with a known or suspected history of intestinal obstruction will be excluded due to the potential risks associated with the administration of bowel preparation agents.
* Known Intolerance to Lactulose or Sodium Phosphate: Participants with a known intolerance to lactulose or sodium phosphate will be excluded due to the risk of severe adverse reactions.
* Pregnancy and Lactation: Pregnant or breastfeeding women will be excluded due to the lack of safety data on bowel preparation agents in this population.
* Interfering Clinical Conditions (Comorbidities): Participants with medical conditions that could interfere with study participation or affect the interpretation of results will be excluded, such as decompensated heart failure, chronic renal or liver disease, and a history of colonic resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale | 1 day
  A total score of 6 or more, with no segment below 2.

SECONDARY OUTCOMES:
Hydroelectrolytic changes. | Two blood drawns: During screening period and baseline visit.
  Number of patients with changes in blood concentrations of sodium, potassium, chloride, creatinine, and urea.
Adverse gastrointestinal effects due to bowel preparation. | Baseline.
  Number of patients experiencing adverse gastrointestinal effects, such as nausea, vomiting, or abdominal distension.
Palatability | Baseline
  Number of patients experiencing changes in taste sensation during bowel preparation intake and its aftertaste: Sweet, salty, bitter, sour. Scale 1-5: low; 5-10: high.
Adenoma detection rate | Baseline
  Quantity and characteristics of adenomas detected during the colonoscopy.

CONTACTS AND LOCATIONS:
Locations (4):
- Mexico (2):
  - Antigüo Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco
  - Nuevo Hospital Civil de Guadalajara "Juan I. Menchaca", Guadalajara, Jalisco
- Panama (2):
  - Hospital Gustavo Nelson Collado Ríos Panamá., Panamá, Herrera Province
  - Hospital Santo Tomas, Bella Vista, Provincia de Panamá

IPD SHARING:
Plan to Share IPD: Undecided
The participants'/patients' data will be recorded only by hospital record and coded ID in the study database, no personal information wil be recorded. If necessary, additional data that may be used in the database will also be considered.